CLINICAL TRIAL: NCT07123974
Title: Implementation Study of a Psychotherapy for Complex Trauma in a French-speaking Setting
Brief Title: Implementing a Therapy for Complex Trauma in French-Speaking Settings
Acronym: TRAUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-3031
Record Dates: First submitted 2025-07-24; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Borderline Personality Disorder (BPD); Complex Post-Traumatic Stress Disorder (CPTSD); Post-Traumatic Stress Disorder, PTSD
Keywords: Psychotherapy research; DBT-PTSD; Mixed-Methods study
MeSH Terms: conditions — Borderline Personality Disorder; Combat Disorders | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dialectical Behaviour Therapy for Post-Traumatic Stress Disorder (DBT-PTSD) (Experimental): Participants receive the Dialectical Behaviour Therapy for Post-Traumatic Stress Disorder (DBT-PTSD) psychotherapy over 45 weekly individual outpatient sessions. All participants followed the same treatment protocol.
  Interventions: Behavioral: Dialectical Behaviour Therapy for Post-Traumatic Stress Disorder (DBT-PTSD)

INTERVENTIONS:
Behavioral: Dialectical Behaviour Therapy for Post-Traumatic Stress Disorder (DBT-PTSD) — DBT-PTSD is 45-week individual psychotherapy (DBT-PTSD) designed to treat adults presenting with both borderline personality disorder (BPD) and complex post-traumatic stress disorder (C-PTSD). The intervention integrates dialectical behavior therapy (DBT) skills, trauma-focused exposure-based interventions, and strategies from compassion-focused therapy and acceptance and commitment therapy. All participants will receive the full sequence of the therapy in outpatient settings, following the structured treatment protocol.

SUMMARY:
Many individuals living with borderline personality disorder (BPD) have experienced childhood trauma, such as abuse or neglect. A significant number of them also meet the criteria for post-traumatic stress disorder (PTSD). However, standard psychotherapies often do not address both conditions at the same time, which can affect treatment outcomes.

A research team in Germany developed and validated a 45-week individual psychotherapy that has shown promising results for individuals coping with both BPD and PTSD. It has already been adapted and offered in English-speaking settings such as Toronto and Boston.

This study aims to adapt this therapy into French in Quebec. Over 24 months, we will conduct a mixed-methods observational study to evaluate changes in symptoms (BPD, PTSD, and other comorbidities) and in daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* PTSD according to the DSM caused by sexual or physical abuse up to the age of 18.
* Three or more criteria for borderline personality disorder (BPD) according to the SCID-II, including affective instability.
* Availability for one year of outpatient treatment (psychotherapy).
* Access to an email address usable for secure links to questionnaires.
* Fluent French-speaking.

Exclusion Criteria:

* Psychotic disorder, bipolar I disorder, intellectual disability, or severe psychopathology requiring immediate care as determined by the treating psychiatrist.
* Severe suicide attempt within two months prior to the inclusion visit.
* Medical condition preventing inclusion (e.g., pregnancy).
* Highly unstable living situation (e.g., homelessness).
* Current substance dependence.
* Having received specific treatment for PTSD or BPD within the year preceding the inclusion visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Patients' qualitative experiences of the treatment | At treatment inclusion, 6-months into treatment and 6-months post-treatment
  Exploration of patients' experiences and perceptions of the treatment through focus groups. No standardized scale or scoring is used. Discussions are audio-recorded, transcribed verbatim, and analyzed thematically to identify common themes related to perceived benefits, challenges, and overall acceptability of the treatment.
Patients' qualitative experiences of the treatment | At treatment initiation, 6-months into treatment and 6-months post-treatment
  Exploration of patients' lived experiences and perceptions of the treatment through semi-structured interviews. No standardized scale or scoring is used. Interviews are transcribed verbatim and thematically analyzed. The outcome focuses on emergent themes related to perceived benefits, challenges, and overall acceptability of the treatment.
Clinicians' qualitative experiences of treatment | At 12 months after treatment initiation and again at 24 months after treatment initiation
  Exploration of therapists' lived experiences and perceptions of the treatment through semi-structured interviews. No standardized scale or scoring is used. Interviews are transcribed verbatim and thematically analyzed. The outcome focuses on emergent themes related to perceived benefits, challenges, and overall acceptability of the treatment.
Participants change in BPD symptom severity | At treatment initiation and every 3 months during the first 12 months of treatment
  The Borderline Symptom List-23 (BSL-23) is a self-report questionnaire consisting of 23 items designed to assess the severity of borderline symptoms. Each item is rated on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("very strong"). The total score is calculated as the mean of all item scores, with a final score that ranges from 0 to 4. Higher scores indicate greater symptom severity.
Participant changes in PTSD symptoms | At treatment initiation and every 3 months during the first 12 months of treatment
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a structured clinical interview used to assess the presence and severity of posttraumatic stress disorder (PTSD) symptoms. It includes 30 items, of which 28 are rated on a 5-point scale ranging from 0 ("absent") to 4 ("extreme/incapacitating"). The total severity score ranges from 0 to 112 (sum of 28 rated items). Higher scores reflect greater PTSD symptom severity.
Participant change in Dissociative experiences | At treatment initiation and every 3 months during the first 12 months of treatment
  Dissociative Experiences Scale (DES) is a 28-item self-report questionnaire designed to assess the frequency of dissociative experiences. Each item is scored as a percentage (0% to 100%) reflecting how often the experience occurs, and the total score corresponds to the mean of all item scores, ranging from 0 to 100. Higher scores indicate more frequent dissociative experiences.
Participant diagnosis of borderline personality disorder | At treatment initation
  Structured Clinical Interview for DSM-IV Axis II Personality Disorders (SCID-II) is a semi-structured diagnostic interview used to assess personality disorders according to DSM-IV criteria. Only standardized questions to assess BPD were used. Each criterion is rated as present, absent, or subthreshold. The interview yields categorical diagnoses rather than a numerical score. A higher score represent a higher severity.
Participant ADHD Screening | At treatment initiation
  Adult ADHD Self-Report Scale (ASRS-v1.1) is an 18-item self-report questionnaire developed to screen for symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) in adults. Part A of the scale consists of 6 items that are most predictive of ADHD. A screening is considered positive if the participant endorses 4 or more items in Part A above the defined threshold. Items are rated on a 5-point Likert scale from 0 ("never") to 4 ("very often"). A positive result suggests the need for further clinical evaluation.
Participant change in depression | At treatment initiation and every 3 months during the first 12 months of treatment
  Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report questionnaire used to assess the severity of depressive symptoms and the presence of suicidal ideation. Each item corresponds to a DSM criterion for major depressive disorder and is rated on a 4-point scale from 0 ("not at all") to 3 ("nearly every day"), yielding a total score ranging from 0 to 27. Higher scores indicate greater depressive symptom severity. Cut-off scores are as follows: 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), and 20-27 (severe depression).
Participant change in suicidal behaviors | At treatment initiation and every 3 months during the first 12 months of treatment
  Suicidal Behaviors Questionnaire-Revised (SBQ-R) is a 4-item self-report questionnaire used to assess risk for suicidal behavior. The items evaluate lifetime suicidal ideation and attempts, frequency of suicidal ideation over the past year, communication of suicidal intent, and self-perceived likelihood of future suicidal behavior. Each item has its own scoring scale, and total scores range from 3 to 18. Higher scores indicate greater risk of suicidal behavior.
Participant alcohol use | At treatment initiation and 12-months into treatment
  Alcohol Use Disorders Identification Test (AUDIT-10) is a 10-item self-report questionnaire developed by the World Health Organization to screen for hazardous and harmful alcohol consumption. Each item is scored from 0 to 4, resulting in a total score ranging from 0 to 40. Higher scores indicate greater severity of alcohol use and associated risk.
Patient impulsivity | At treatment initiation and 12-months into treatment
  UPPS-P Impulsive Behavior Scale is a self-report questionnaire designed to assess five distinct facets of impulsivity: Negative Urgency, Lack of Premeditation, Lack of Perseverance, Sensation Seeking, and Positive Urgency. The full version includes 59 items rated on a 4-point Likert scale from 1 ("agree strongly") to 4 ("disagree strongly"), with subscale scores and a total score calculated by summing relevant items. Higher scores reflect greater levels of impulsive traits.
Participant and Clinician Working Alliance | Every 3 months during the first 12 months of treatment
  Working Alliance Inventory - Short Form (WAI-SF) is a 12-item self-report questionnaire that assesses the quality of the therapeutic alliance between a client and therapist. Each item is rated on a 7-point Likert scale from 1 ("never") to 7 ("always"), yielding a total score ranging from 12 to 84. Higher scores indicate a stronger perceived working alliance.
Clinician treatment adherence to DBT-PTSD | Two sessions per therapist, scheduled at random points during the 12-month treatment period
  Adherence Rating Scale for DBT-PTSD (ARS-DBT-PTSD) is a clinician-rated instrument designed to assess therapist adherence to the Dialectical Behavior Therapy protocol adapted for Posttraumatic Stress Disorder (DBT-PTSD). The scale includes a structured set of items evaluating specific therapeutic strategies, techniques, and session structure elements, each rated on a standardized scale (typically from 0 = "not implemented" to 2 or 3 = "fully implemented"). Higher scores reflect greater adherence to the DBT-PTSD treatment model.
Clinician competence for DBT-PTSD | Two sessions per therapist, scheduled at random points during the 12-month treatment period
  Competence Rating Scale for DBT-PTSD is a clinician-rated instrument designed to assess the therapist's competence in delivering Dialectical Behavior Therapy adapted for Posttraumatic Stress Disorder (DBT-PTSD). It evaluates the quality of therapeutic delivery across several domains, such as treatment structure, application of DBT principles, interpersonal effectiveness, and responsiveness to trauma-related content. Each item is typically rated on a Likert-type scale (e.g., from 0 = "inadequate" to 6 = "excellent"). Higher scores indicate greater therapist competence in applying the DBT-PTSD model.
Participant change in functioning | At treatment initiation and every 3 months during the first 12 months of treatment
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) is a standardized self-report questionnaire developed by the WHO to assess disability and functional impairment across six domains: cognition, mobility, self-care, getting along, life activities, and participation. The 36-item version rates each item on a 5-point Likert scale from 1 ("none") to 5 ("extreme or cannot do"), with total scores ranging from 36 to 180. Scores can be summed or converted into a standardized score from 0 to 100, where higher scores reflect greater disability and functional impairment.
Participant ADHD Screening | At treatment initiation
  Wender Utah Rating Scale (WURS) is a 50-item self-report questionnaire used to retrospectively assess symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) in childhood. Each item is rated on a 5-point Likert scale from 0 ("not at all or never") to 4 ("very much or very often"), yielding a total score ranging from 0 to 200. A total score of 51 or higher is considered indicative of possible childhood ADHD.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Cailhol, Principal Investigator — Ciusss de l'Est de Montréal, Université de Montréal
Locations (1):
- Institut universitaire en santé mentale de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No